CLINICAL TRIAL: NCT00814307
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Of The Efficacy And Safety Of 2 Doses Of CP-690,550 Monotherapy In Patients With Active Rheumatoid Arthritis
Brief Title: A Phase 3 Study Comparing 2 Doses of CP-690,550 vs. Placebo for Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921045
Record Dates: First submitted 2008-12-22; First posted 2008-12-24 (Estimated); Results first posted 2013-01-11 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: Antirheumatic Agents Clinical Trial
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active 5mg (Experimental)
  Interventions: Drug: CP-690,550
- Active 10 mg (Experimental)
  Interventions: Drug: CP-690,550
- Placebo Sequence 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo Sequence 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CP-690,550 — 5mg CP-690,550 BID PO for 6 months
  Arms: Active 5mg
Drug: CP-690,550 — 10 mg CP-690,550 BID PO for 6 months
  Arms: Active 10 mg
Drug: Placebo — Placebo patients advance to 5mg CP-690,550 BID at Month 3 visit
  Arms: Placebo Sequence 1
Drug: Placebo — Placebo patients advance to 10mg CP-690,550 BID at Month 3 visit
  Arms: Placebo Sequence 2

SUMMARY:
This Phase 3 study is intended to provide evidence of the efficacy and safety of CP 690,550 when dosed 5 mg and 10 mg twice a day as monotherapy in adult patients with moderate to severe Rheumatoid Arthritis. It is intended to confirm the benefits of CP-690,550 in improving signs and symptoms and physical function that were observed in the Phase 2 Rheumatoid Arthritis studies.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of RA based upon the American College of Rheumatology (ACR) 1987 Revised Criteria.
* The patient has active disease at both Screening and Baseline, as defined by both: ≥6 joints tender or painful on motion; and ≥6 joints swollen; and fulfills 1 of the following 2 criteria at Screening: 1.ESR (Westergren method) >28 mm in the local laboratory. 2. CRP >7 mg/L in the central laboratory
* Patient had an inadequate response to at least one DMARD (traditional or biologic) due to lack of efficacy or toxicity.
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis.
* Patient has washed out of all DMARDs other that antimalarials

Exclusion Criteria:

* Blood dyscrasias including confirmed: 1. Hemoglobin <9 g/dL or Hematocrit <30%; 2. White blood cell count <3.0 x 109/L; 3. Absolute neutrophil count <1.2 x 109/L; 4. Platelet count <100 x 109/L
* History of any other autoimmune rheumatic disease other than Sjogren's syndrome
* No malignancy or history of malignancy.
* History of infection requiring hospitalization, parenteral antimicrobial therapy, or as otherwise judged clinically significant by the investigator, within the 6 months prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (83):
- United States (30):
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Venice, Florida
  - Pfizer Investigational Site, Zephyrhills, Florida
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Hyannis, Massachusetts
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Teaneck, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Olean, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Rocky Mount, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Mesquite, Texas
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Clarksburg, West Virginia
- Brazil (5):
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Bulgaria (3):
  - Pfizer Investigational Site, Pleven
  - Pfizer Investigational Site, Plovdiv
  - Pfizer Investigational Site, Sofia
- Chile (2):
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Providencia, Santiago, RM
- Colombia (2):
  - Pfizer Investigational Site, Bucaramanga, Santander Department
  - Pfizer Investigational Site, Barranquilla
- Czechia (6):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Česká Lípa
  - Pfizer Investigational Site, Hlučín
  - Pfizer Investigational Site, Pardubice
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Zlín
- Pfizer Investigational Site, Santo Domingo, Santo Domingo Province, Dominican Republic
- Germany (6):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Nuremberg
- India (6):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Secunderabad, Andhra Pradesh
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mangalore, Karnataka
  - Pfizer Investigational Site, Pune, Maharashtra
- Malaysia (4):
  - Pfizer Investigational Site, Putrajaya, Kuala Lumpur
  - Pfizer Investigational Site, Kota Kinabalu, Sabah
  - Pfizer Investigational Site, Kuching, Sarawak
  - Pfizer Investigational Site, Petaling Jaya, Selangor
- Mexico (4):
  - Pfizer Investigational Site, Chihuahua City, Chihuahua
  - Pfizer Investigational Site, Tijuana, Estado de Baja California
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Philippines (4):
  - Pfizer Investigational Site, Dasmariñas, Cavite
  - Pfizer Investigational Site, Bajada, Davao City, Phlippines
  - Pfizer Investigational Site, Las Piñas
  - Pfizer Investigational Site, Manila
- Poland (2):
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Pfizer Investigational Site, San Juan, Puerto Rico
- Russia (2):
  - Pfizer Investigational Site, Petrozavodsk
  - Pfizer Investigational Site, Smolensk
- Ukraine (5):
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Simferopol, Crimea
  - Pfizer Investigational Site, Vinnitsa

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Pope J, Finckh A, Silva-Fernandez L, Mandl P, Fan H, Rivas JL, Valderrama M, Montoro M. Tofacitinib Monotherapy in Rheumatoid Arthritis: Clinical Trials and Real-World Data Contextualization of Patients, Efficacy, and Treatment Retention. Open Access Rheumatol. 2024 Jun 11;16:115-126. doi: 10.2147/OARRR.S446431. eCollection 2024. PMID 38883150
- [Derived] Citera G, Jain R, Irazoque F, Madariaga H, Gruben D, Wang L, Stockert L, Santana K, Ebrahim A, Ponce de Leon D. Tofacitinib Efficacy in Patients with Rheumatoid Arthritis and Probable Depression/Anxiety: Post Hoc Analysis of Phase 3 and 3b/4 Randomized Controlled Trials. Rheumatol Ther. 2024 Feb;11(1):35-50. doi: 10.1007/s40744-023-00612-7. Epub 2023 Nov 5. PMID 37925660
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Dougados M, Taylor PC, Bingham CO 3rd, Fallon L, Brault Y, Roychoudhury S, Wang L, Kessouri M. The effect of tofacitinib on residual pain in patients with rheumatoid arthritis and psoriatic arthritis. RMD Open. 2022 Sep;8(2):e002478. doi: 10.1136/rmdopen-2022-002478. PMID 36814062
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Dikranian AH, Gonzalez-Gay MA, Wellborne F, Alvaro-Gracia JM, Takiya L, Stockert L, Paulissen J, Shi H, Tatulych S, Curtis JR. Efficacy of tofacitinib in patients with rheumatoid arthritis stratified by baseline body mass index: an analysis of pooled data from phase 3 studies. RMD Open. 2022 May;8(1):e002103. doi: 10.1136/rmdopen-2021-002103. PMID 35577477
- [Derived] Dikranian A, Gold D, Bessette L, Nash P, Azevedo VF, Wang L, Woolcott J, Shapiro AB, Szumski A, Fleishaker D, Wollenhaupt J. Frequency and Duration of Early Non-serious Adverse Events in Patients with Rheumatoid Arthritis and Psoriatic Arthritis Treated with Tofacitinib. Rheumatol Ther. 2022 Apr;9(2):411-433. doi: 10.1007/s40744-021-00405-w. Epub 2021 Dec 17. PMID 34921355
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Kivitz AJ, Cohen S, Keystone E, van Vollenhoven RF, Haraoui B, Kaine J, Fan H, Connell CA, Bananis E, Takiya L, Fleischmann R. A pooled analysis of the safety of tofacitinib as monotherapy or in combination with background conventional synthetic disease-modifying antirheumatic drugs in a Phase 3 rheumatoid arthritis population. Semin Arthritis Rheum. 2018 Dec;48(3):406-415. doi: 10.1016/j.semarthrit.2018.07.006. Epub 2018 Jul 19. PMID 30177460
- [Derived] Bird P, Bensen W, El-Zorkany B, Kaine J, Manapat-Reyes BH, Pascual-Ramos V, Witcombe D, Soma K, Zhang R, Thirunavukkarasu K. Tofacitinib 5 mg Twice Daily in Patients with Rheumatoid Arthritis and Inadequate Response to Disease-Modifying Antirheumatic Drugs: A Comprehensive Review of Phase 3 Efficacy and Safety. J Clin Rheumatol. 2019 Apr;25(3):115-126. doi: 10.1097/RHU.0000000000000786. PMID 29794874
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Strand V, Kremer J, Wallenstein G, Kanik KS, Connell C, Gruben D, Zwillich SH, Fleischmann R. Effects of tofacitinib monotherapy on patient-reported outcomes in a randomized phase 3 study of patients with active rheumatoid arthritis and inadequate responses to DMARDs. Arthritis Res Ther. 2015 Nov 4;17:307. doi: 10.1186/s13075-015-0825-9. PMID 26530039
- [Derived] Charles-Schoeman C, Burmester G, Nash P, Zerbini CA, Soma K, Kwok K, Hendrikx T, Bananis E, Fleischmann R. Efficacy and safety of tofacitinib following inadequate response to conventional synthetic or biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2016 Jul;75(7):1293-301. doi: 10.1136/annrheumdis-2014-207178. Epub 2015 Aug 14. PMID 26275429
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- [Derived] Fleischmann R, Kremer J, Cush J, Schulze-Koops H, Connell CA, Bradley JD, Gruben D, Wallenstein GV, Zwillich SH, Kanik KS; ORAL Solo Investigators. Placebo-controlled trial of tofacitinib monotherapy in rheumatoid arthritis. N Engl J Med. 2012 Aug 9;367(6):495-507. doi: 10.1056/NEJMoa1109071. PMID 22873530
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921045&StudyName=A%20Phase%203%20study%20comparing%202%20doses%20of%20CP-690%2C550%20vs.%20placebo%20for%20treatment%20of%20rheumatoid%20arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 5 mg: CP-690,550 5 milligram (mg) tablet orally twice daily up to Month 6.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily up to Month 6.
- Placebo, Then CP-690,550 5 mg: Matching placebo tablet orally twice daily up to Month 3 followed by CP-690,550 5 mg tablet twice daily from Month 3 up to Month 6 or early termination.
- Placebo, Then CP-690,550 10 mg: Matching placebo tablet orally twice daily up to Month 3 followed by CP-690,550 10 mg tablet twice daily from Month 3 up to Month 6 or early termination.
Period: Overall Study
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Started | 244 | 245 | 61 | 61
Treated | 243 | 245 | 61 | 61
Completed | 232 | 218 | 54 | 51
Not Completed | 12 | 27 | 7 | 10
Not completed — Randomized but not treated | 1 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 9 | 3 | 2
Not completed — Lack of Efficacy | 1 | 1 | 3 | 4
Not completed — Other | 1 | 2 | 0 | 1
Not completed — Protocol Violation | 2 | 8 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 6 | 0 | 2
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Total
Number analyzed (Participants) | 243 | 245 | 61 | 61 | 610
Age Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (11.5) | 52.4 (11.7) | 50.7 (12.8) | 48.8 (11.9) | 51.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 216 | 54 | 51 | 528
  Male | 36 | 29 | 7 | 10 | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Month 3
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Month 3
Population: Full Analysis Set (FAS): all randomized participants who received at least 1 dose of study drug (CP-690550/placebo), had at least 1 post-baseline measurement, and baseline measurement for change from baseline endpoint. 'N' (number of participants analyzed)=participants evaluable for this measure.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Matching placebo tablet orally twice daily up to Month 3.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 241 | 242 | 120
percentage of participants | 59.75 | 65.70 | 26.67
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Normal approximation for the difference in binomial proportions was used to test the superiority of each dose of CP-690,550 to placebo; Test type: Superiority or Other; p < 0.0001, Normal approximation — A step-down procedure was used to control for multiple comparisons. In order for the comparison to 5 mg to be statistically significant, the comparison to 10 mg had to be statistically significant; Percent difference = 39.04, 95% CI 2-sided [29.12 to 48.95]
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Normal approximation — [p-value comment as in outcome 1, analysis 1]; Percent difference = 33.08, 95% CI 2-sided [23.04 to 43.13]

2. Primary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Month 3
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 functional categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3, 0=least functional difficulty and 3=extreme functional difficulty.
Time Frame: Baseline, Month 3
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 240 | 241 | 122
units on a scale
  Baseline (n=240,241,122) | 1.53 (0.66) | 1.50 (0.64) | 1.53 (0.65)
  Change at Month 3 (n=237,227,109) | -0.48 (0.66) | -0.54 (0.60) | -0.18 (0.61)
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; p-value was calculated using linear mixed effect model. The fixed effects of treatment, visit, and treatment-by-visit interaction were included, along with participant as random effect; Test type: Superiority or Other; p < .0001, Linear mixed effect model — A step-down procedure was used to control for multiple comparisons. For comparison of 10 mg to placebo to be statistically significant in this measure, comparison of 10 mg to placebo in ACR20 had to be significant; Least squares mean difference = -0.38, 95% CI 2-sided [-0.50 to -0.27]
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Linear mixed effect model — A step-down procedure was used to control for multiple comparisons. For comparison of 5 mg to placebo to be statistically significant, comparison of 10 mg to placebo and comparison of 5 mg to placebo in ACR20 had to be statistically significant; Least squares mean difference = -0.31, 95% CI 2-sided [-0.43 to -0.20]

3. Primary Outcome: Percentage of Participant With Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than 2.6 at Month 3
Description: DAS28-4 (ESR) calculated from swollen joint count (SJC) and tender/painful joint count (TJC) using 28 joint count, erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PtGA) of disease activity (transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) less than or equal to (=<) 3.2 implied low disease activity, greater than (>) 3.2 to 5.1 implied moderate to high disease activity and less than (<) 2.6=remission.
Time Frame: Month 3
Population: FAS: all participants who were randomized to study, received at least 1 dose of study drug (CP-690550/placebo), had at least 1 post-baseline measurement, and baseline measurement for change from baseline endpoint. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 229 | 219 | 104
percentage of participants | 6.11 | 10.05 | 4.81
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Normal approximation for the difference in binomial proportions was used to test the superiority of each dose of CP-690550 to placebo; Test type: Superiority or Other; p = 0.0728, Normal Approximation — A step-down procedure was used to control for multiple comparisons. For comparison of 10 mg to placebo to be statistically significant in this measure, comparison of 10 mg to placebo in HAQ-DI had to be significant; Percent difference = 5.24, 95% CI 2-sided [-0.49 to 10.96]
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.6193, Normal Approximation — A step-down procedure was used to control for multiple comparisons. For comparison of 5 mg to placebo to be statistically significant, comparison of 10 mg to placebo and comparison of 5 mg to placebo in HAQ-DI had to be statistically significant; Percent difference = 1.31, 95% CI 2-sided [-3.85 to 6.46]

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 2, Month 1 and 2
Description: ACR20 response: >= 20% improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 2, Month 1, 2
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 241 | 242 | 120
percentage of participants
  Week 2 | 29.58 | 39.17 | 11.76
  Month 1 | 46.47 | 52.07 | 21.67
  Month 2 | 56.85 | 60.74 | 25.83

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Month 4, 5 and 6
Description: as for outcome 4
Time Frame: Month 4, 5, 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 241 | 242 | 60 | 60
percentage of participants
  Month 4 | 69.29 | 69.01 | 51.67 | 61.67
  Month 5 | 68.46 | 69.83 | 61.67 | 63.33
  Month 6 | 69.29 | 71.07 | 58.33 | 56.67

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Week 2, Month 1, 2 and 3
Description: ACR50 response: greater than or equal to >=50% improvement in tender joint count; >=50% improvement in swollen joint count; and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Week 2, Month 1, 2, 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 241 | 242 | 120
percentage of participants
  Week 2 | 5.83 | 12.92 | 4.20
  Month 1 | 17.43 | 23.97 | 4.17
  Month 2 | 26.14 | 33.88 | 5.83
  Month 3 | 31.12 | 36.78 | 12.50

7. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Month 4, 5 and 6
Description: as for outcome 6
Time Frame: Month 4, 5, 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 241 | 242 | 60 | 60
percentage of participants
  Month 4 | 37.34 | 42.98 | 28.33 | 28.33
  Month 5 | 39.42 | 45.45 | 36.67 | 35.00
  Month 6 | 41.91 | 46.69 | 33.33 | 33.33

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Week 2, Month 1, 2 and 3
Description: ACR70 response: >=70% improvement in tender joint count; >=70% improvement in swollen joint count; and >=70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of HAQ); and CRP.
Time Frame: Week 2, Month 1, 2, 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 241 | 242 | 120
percentage of participants
  Week 2 | 2.08 | 4.58 | 0.00
  Month 1 | 4.98 | 9.09 | 1.67
  Month 2 | 9.96 | 19.01 | 3.33
  Month 3 | 15.35 | 20.25 | 5.83

9. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Month 4, 5 and 6
Description: as for outcome 8
Time Frame: Month 4, 5, 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 241 | 242 | 60 | 60
percentage of participants
  Month 4 | 19.92 | 26.03 | 13.33 | 15.00
  Month 5 | 21.16 | 28.51 | 18.33 | 18.33
  Month 6 | 21.99 | 29.34 | 20.00 | 21.67

10. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Baseline and Month 3
Description: DAS28-4 (ESR) calculated from SJC and TJC using 28 joint count, ESR (mm/hour) and PtGA of disease activity (transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Month 3
Population: FAS population. 'N' (number of participants analyzed)=participants evaluable for this measure. 'n'=participants evaluable at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 236 | 234 | 115
units on a scale
  Baseline (n= 236, 234, 115) | 6.71 (0.93) | 6.70 (0.94) | 6.65 (0.93)
  Month 3 (n= 229, 219, 104) | 4.78 (1.37) | 4.55 (1.39) | 5.54 (1.46)

11. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Month 6
Description: as for outcome 3
Time Frame: Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 221 | 209 | 52 | 47
units on a scale | 4.33 (1.39) | 4.01 (1.38) | 4.31 (1.34) | 3.98 (1.50)

12. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Baseline, Week 2, Month 1, 2 and 3
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (milligram per liter [mg/L]). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Week 2, Month 1, 2, 3
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n'=participants evaluable at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 239 | 242 | 121
units on a scale
  Baseline (n= 239, 242, 121) | 5.68 (0.90) | 5.60 (0.91) | 5.56 (0.85)
  Week 2 (n= 234, 231, 118) | 4.79 (1.12) | 4.42 (1.11) | 5.30 (1.13)
  Month 1 (n= 237, 236, 115) | 4.41 (1.12) | 3.99 (1.26) | 4.98 (1.25)
  Month 2 (n= 238, 233, 109) | 4.02 (1.26) | 3.64 (1.27) | 4.85 (1.36)
  Month 3 (n= 238, 229, 109) | 3.89 (1.27) | 3.59 (1.27) | 4.68 (1.27)

13. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Month 4, 5 and 6
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Month 4, 5, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 235 | 222 | 55 | 50
units on a scale
  Month 4 (n= 235, 222, 54, 48) | 3.65 (1.24) | 3.26 (1.22) | 3.89 (1.19) | 3.50 (1.28)
  Month 5 (n= 231, 219, 55, 50) | 3.54 (1.26) | 3.12 (1.24) | 3.53 (1.25) | 3.34 (1.26)
  Month 6 (n= 228, 215, 53, 50) | 3.48 (1.23) | 3.11 (1.26) | 3.56 (1.32) | 3.12 (1.34)

14. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) at Baseline, Week 2, Month 1, 2 and 3
Description: as for outcome 2
Time Frame: Baseline, Week 2, Month 1, 2, 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 240 | 241 | 122
units on a scale
  Baseline (n= 240, 241, 122) | 1.53 (0.66) | 1.50 (0.64) | 1.53 (0.65)
  Week 2 (n= 240, 239, 119) | 1.27 (0.62) | 1.21 (0.65) | 1.43 (0.64)
  Month 1 (n= 237, 240, 116) | 1.18 (0.68) | 1.09 (0.66) | 1.40 (0.64)
  Month 2 (n= 240, 233, 110) | 1.05 (0.66) | 0.97 (0.68) | 1.40 (0.68)
  Month 3 (n= 238, 229, 109) | 1.05 (0.70) | 0.97 (0.69) | 1.35 (0.73)

15. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) at Month 4, 5 and 6
Description: as for outcome 2
Time Frame: Month 4, 5, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 235 | 223 | 55 | 50
units on a scale
  Month 4 (n= 235, 223, 55, 49) | 0.97 (0.66) | 0.88 (0.68) | 1.08 (0.70) | 1.09 (0.65)
  Month 5 (n= 231, 221, 55, 50) | 0.95 (0.69) | 0.87 (0.69) | 1.04 (0.59) | 1.03 (0.64)
  Month 6 (n= 229, 216, 54, 50) | 0.94 (0.68) | 0.86 (0.67) | 1.05 (0.63) | 1.00 (0.66)

16. Secondary Outcome: Patient Assessment of Arthritis Pain at Baseline, Week 2, Month 1, 2 and 3
Description: Participants assessed the severity of their arthritis pain using a 100 millimeter (mm) visual analog scale (VAS). The scale ranged from 0 (no pain) to 100 (most severe pain), measurement on a scale corresponds to the magnitude of their pain.
Time Frame: Baseline, Week 2, Month 1, 2, 3
Population: FAS: all participants who were randomized to study, received at least 1 dose of study drug (CP-690550/placebo), had at least 1 post-baseline measurement, and baseline measurement for change from baseline endpoint. 'n'=participants evaluable at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 241 | 243 | 122
mm
  Baseline (n= 241, 243, 122) | 61.35 (22.27) | 62.03 (23.63) | 61.79 (21.27)
  Week 2 (n= 239, 239, 119) | 45.92 (22.87) | 42.13 (25.06) | 55.61 (23.63)
  Month 1 (n= 237, 240, 116) | 40.68 (23.04) | 36.86 (24.46) | 52.47 (24.59)
  Month 2 (n= 240, 233, 110) | 36.39 (23.29) | 31.66 (24.38) | 52.38 (26.09)
  Month 3 (n= 237, 228, 108) | 34.93 (23.73) | 31.37 (24.35) | 49.84 (25.10)

17. Secondary Outcome: Patient Assessment of Arthritis Pain at Month 4, 5 and 6
Description: Participants assessed the severity of their arthritis pain using a 100 mm visual analog scale (VAS). The scale ranged from 0 (no pain) to 100 (most severe pain), measurement on a scale corresponds to the magnitude of their pain.
Time Frame: Month 4, 5, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 235 | 223 | 55 | 50
mm
  Month 4 (n= 235, 223, 55, 49) | 33.18 (23.02) | 29.70 (23.21) | 34.27 (24.53) | 35.47 (25.28)
  Month 5 (n= 231, 221, 55, 50) | 32.63 (23.07) | 29.10 (22.24) | 34.05 (23.48) | 35.06 (24.82)
  Month 6 (n= 228, 216, 54, 50) | 32.60 (23.55) | 27.89 (23.17) | 33.96 (24.62) | 32.28 (23.79)

18. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain at Baseline, Week 2, Month 1, 2 and 3
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm Visual Analog Scale where 0 = very well and 100 = very poorly.
Time Frame: Baseline, Week 2, Month 1, 2, 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 240 | 243 | 122
mm
  Baseline (n= 240, 243, 122) | 61.66 (22.00) | 63.46 (23.23) | 62.63 (21.91)
  Week 2 (n= 240, 239, 119) | 46.34 (22.36) | 41.32 (24.90) | 55.95 (23.79)
  Month 1 (n= 237, 240, 116) | 39.63 (22.36) | 37.69 (23.94) | 53.23 (24.01)
  Month 2 (n= 240, 233, 110) | 36.29 (22.20) | 32.56 (23.47) | 53.05 (26.04)
  Month 3 (n= 238, 229, 108) | 35.90 (23.61) | 32.78 (23.75) | 50.48 (25.82)

19. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain at Month 4, 5 and 6
Description: as for outcome 18
Time Frame: Month 4, 5, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 235 | 223 | 55 | 50
mm
  Month 4 (n= 235, 223, 55, 49) | 33.59 (22.44) | 29.69 (22.25) | 35.27 (23.77) | 36.45 (25.92)
  Month 5 (n= 231, 221, 55, 50) | 34.59 (23.37) | 29.37 (22.13) | 32.88 (21.43) | 33.96 (25.02)
  Month 6 (n= 228, 216, 54, 50) | 32.56 (23.09) | 29.52 (22.89) | 33.51 (24.00) | 32.89 (23.78)

20. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis Pain at Baseline, Week 2, Month 1, 2 and 3
Description: Physician Global Assessment of Arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: Baseline, Week 2, Month 1, 2, 3
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 241 | 243 | 122
mm
  Baseline (n= 241, 243, 122) | 61.46 (16.93) | 60.84 (16.84) | 62.22 (16.85)
  Week 2 (n= 239, 240, 119) | 43.43 (17.69) | 40.47 (19.73) | 52.15 (19.25)
  Month 1 (n= 237, 240, 116) | 35.89 (18.91) | 33.99 (20.37) | 46.98 (22.29)
  Month 2 (n= 240, 232, 110) | 32.06 (20.81) | 26.75 (19.23) | 44.45 (23.62)
  Month 3 (n= 238, 229, 109) | 29.20 (19.98) | 24.47 (18.42) | 42.05 (23.58)

21. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis Pain at Month 4, 5 and 6
Description: as for outcome 20
Time Frame: Month 4, 5, 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 235 | 221 | 55 | 50
mm
  Month 4 (n= 235, 221, 54, 49) | 25.30 (18.56) | 21.21 (16.46) | 27.48 (19.80) | 25.86 (20.32)
  Month 5 (n= 231, 221, 55, 50) | 23.60 (17.63) | 20.99 (16.13) | 24.74 (17.93) | 25.90 (19.85)
  Month 6 (n= 229, 216, 54, 50) | 23.26 (18.12) | 20.61 (16.27) | 26.16 (19.55) | 21.54 (17.51)

22. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) at Baseline, Month 3
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning) and is reported as 2 summary scores; Physical Component Score and Mental Component Score. Total score range for the summary scores = 0- 100, where higher score represents higher level of functioning.
Time Frame: Baseline, Month 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 239 | 243 | 122
units on a scale
  Baseline:Physical functioning (n=239,243,122) | 30.09 (9.31) | 30.51 (8.76) | 31.41 (9.66)
  Baseline:Role Physical (n=239,243,122) | 32.84 (8.87) | 33.45 (8.69) | 33.33 (8.97)
  Baseline:Social Functioning (n=239,243,122) | 36.78 (11.04) | 36.07 (11.27) | 35.16 (10.34)
  Baseline:Bodily Pain (n=239,243,122) | 32.41 (7.57) | 32.74 (7.55) | 32.77 (7.67)
  Baseline:Mental Health (n=239,243,122) | 40.05 (11.49) | 40.50 (12.57) | 38.43 (12.36)
  Baseline:Role Emotional (n=239,243,122) | 34.26 (12.63) | 36.70 (13.03) | 35.17 (13.11)
  Baseline:Vitality (n=239,243,122) | 41.22 (10.06) | 41.04 (10.27) | 40.13 (9.82)
  Baseline:General health perception(n=239,243,122) | 34.86 (8.72) | 35.71 (8.86) | 34.70 (9.00)
  Baseline:Mental Component (n=239,243,122) | 41.36 (11.68) | 42.19 (12.44) | 39.87 (11.62)
  Baseline:Physical Component (n=239,243,122) | 31.23 (8.03) | 31.37 (7.39) | 32.21 (8.35)
  Month 3:Physical functioning(n=235,224,108) | 36.13 (10.44) | 37.05 (10.58) | 32.93 (10.63)
  Month 3:Role Physical (n=233,224,107) | 38.90 (9.41) | 40.45 (9.90) | 35.19 (9.72)
  Month 3:Social Functioning(n=235,224,108) | 41.62 (10.90) | 43.25 (9.95) | 36.14 (10.04)
  Month 3:Bodily Pain (n=235,224,108) | 40.56 (9.38) | 43.08 (9.50) | 36.35 (8.81)
  Month 3:Mental Health (n=235,224,108) | 44.33 (11.50) | 45.13 (11.25) | 40.73 (10.73)
  Month 3:Role Emotional (n=233,224,107) | 38.76 (12.13) | 40.84 (11.57) | 36.08 (12.66)
  Month 3:Vitality (n=235,224,108) | 47.36 (10.69) | 49.03 (9.86) | 42.23 (9.75)
  Month 3:General health perception(n=235,224,108) | 39.52 (9.37) | 41.50 (9.78) | 37.22 (8.75)
  Month 3:Mental Component (n=233,224,107) | 45.21 (11.65) | 46.58 (10.81) | 41.13 (10.90)
  Month 3:Physical Component (n=233,224,107) | 38.03 (9.18) | 39.69 (9.31) | 34.58 (8.94)

23. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) at Month 6
Description: as for outcome 22
Time Frame: Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 229 | 216 | 54 | 50
units on a scale
  Physical functioning | 36.99 (10.07) | 38.43 (10.67) | 35.74 (10.23) | 35.26 (9.98)
  Role Physical | 39.85 (9.57) | 40.93 (9.50) | 38.25 (9.73) | 38.97 (9.06)
  Social Functioning | 42.36 (10.60) | 42.98 (10.15) | 39.57 (11.45) | 43.39 (9.78)
  Bodily Pain | 41.80 (9.55) | 43.67 (9.54) | 40.80 (9.36) | 42.19 (9.46)
  Mental Health | 43.98 (12.18) | 45.05 (11.01) | 42.14 (11.90) | 47.03 (10.62)
  Role Emotional | 40.37 (11.32) | 41.03 (11.47) | 39.04 (12.93) | 42.66 (12.10)
  Vitality | 47.47 (10.58) | 48.89 (10.29) | 45.08 (9.50) | 47.88 (9.19)
  General health perception | 41.05 (9.24) | 42.58 (9.84) | 38.99 (8.73) | 40.42 (10.83)
  Mental component | 45.43 (11.58) | 46.08 (10.44) | 43.29 (12.37) | 48.76 (11.06)
  Physical component | 39.24 (8.42) | 40.89 (9.04) | 37.89 (9.56) | 37.06 (9.14)

24. Secondary Outcome: Medical Outcome Study Sleep Scale (MOS-SS) at Baseline and Month 3
Description: Participant-rated 12 item questionnaire assess constructs of sleep over past week.7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence (range:0-100); sleep quantity(range:0-24), optimal sleep(yes or no). 9 item index measures of sleep disturbance provide composite scores: sleep problem summary, overall sleep problem. Except Adequacy, Optimal, Quantity of sleep, higher scores=more impairment. Scores transformed(actual raw score minus lowest possible score divided by possible raw score range*100);total score range:0-100,higher score=more intensity of attribute.
Time Frame: Baseline, Month 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 239 | 242 | 122
units on a scale
  Baseline:overall sleep problem(n=238,242,122) | 42.45 (18.38) | 43.09 (20.41) | 47.32 (21.24)
  Baseline:sleep problem summary(n=239,242,122) | 40.59 (18.98) | 42.38 (21.01) | 45.98 (21.85)
  Baseline:somnolence(n=239,243,122) | 37.21 (22.47) | 37.64 (21.76) | 36.56 (21.29)
  Baseline:snoring(n=238,243,121) | 35.71 (31.07) | 30.29 (30.50) | 30.25 (31.42)
  Baseline:quantity(n=240,243,122) | 6.53 (1.56) | 6.38 (1.63) | 6.37 (1.74)
  Baseline:sleep disturbance(n=238,242,122) | 44.44 (24.11) | 43.33 (26.18) | 51.27 (25.89)
  Baseline:awaken short of breath(n=239,243,122) | 18.16 (23.76) | 20.91 (25.47) | 24.92 (29.35)
  Baseline:adequacy(n=239,243,122) | 45.44 (27.25) | 42.63 (27.37) | 40.08 (28.36)
  Month 3:overall sleep problem(n=236,228,109) | 35.53 (19.30) | 33.29 (19.96) | 41.13 (21.31)
  Month 3:sleep problem summary(n=236,228,109) | 34.46 (19.89) | 33.25 (20.16) | 40.55 (22.02)
  Month 3:somnolence(n=236,229,109) | 30.28 (21.28) | 30.45 (21.26) | 35.66 (23.01)
  Month 3:snoring(n=236,229,109) | 32.63 (29.61) | 25.85 (27.57) | 27.52 (29.79)
  Month 3:quantity(n=237,228,109) | 6.77 (1.63) | 6.89 (1.45) | 6.78 (1.47)
  Month 3:sleep disturbance(n=236,229,109) | 36.58 (24.67) | 32.58 (24.27) | 41.16 (27.40)
  Month 3:awaken short of breath(n=236,228,109) | 15.93 (21.29) | 16.23 (21.69) | 22.20 (24.99)
  Month 3:adequacy(n=236,229,109) | 51.69 (28.77) | 52.93 (27.75) | 44.40 (27.67)

25. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study Sleep Scale (MOS-SS) at Baseline and Month 3
Description: MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence, sleep quantity and optimal sleep. Participants responded whether their sleep was optimal or not by choosing yes or no. Number of participants with optimal sleep are reported.
Time Frame: Baseline, Month 3
Population: FAS population. 'n'=participants evaluable at given time point for each group respectively.
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 241 | 243 | 122
participants
  Baseline(n=241,243,122) | 96 | 98 | 45
  Month 3(n=238,229,109) | 113 | 117 | 52

26. Secondary Outcome: Medical Outcome Study Sleep Scale (MOS-SS) at Month 6
Description: as for outcome 24
Time Frame: Month 6
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 229 | 214 | 54 | 50
units on a scale
  Overall sleep problem | 35.68 (18.80) | 33.33 (19.19) | 37.29 (19.26) | 35.64 (21.20)
  Sleep problem summary | 35.17 (18.81) | 33.33 (19.66) | 37.41 (20.30) | 35.87 (20.80)
  Somnolence | 30.26 (21.01) | 29.42 (20.64) | 31.36 (19.75) | 29.60 (21.56)
  Snoring | 35.28 (31.04) | 27.79 (28.24) | 26.30 (28.50) | 29.20 (27.47)
  Quantity | 6.64 (1.45) | 6.87 (1.71) | 6.65 (1.52) | 6.64 (1.27)
  Sleep disturbance | 35.75 (25.11) | 33.38 (23.91) | 37.80 (23.96) | 33.80 (25.83)
  Awaken short of breath | 15.55 (21.67) | 15.70 (21.41) | 21.11 (21.43) | 23.20 (25.67)
  Adequacy(n=229,214,54,50) | 48.52 (27.41) | 53.04 (29.14) | 49.44 (29.36) | 49.00 (27.94)

27. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study Sleep Scale (MOS-SS) at Month 6
Description: as for outcome 25
Time Frame: Month 6
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 229 | 216 | 54 | 50
participants | 105 | 107 | 23 | 25

28. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale at Baseline and Month 3
Description: FACIT-Fatigue is a 13-item questionnaire. Participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Month 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 240 | 243 | 122
units on a scale
  Baseline (n= 240, 243, 122) | 27.90 (10.70) | 27.72 (11.15) | 27.17 (10.88)
  Month 3 (n= 237, 227, 109) | 34.40 (10.65) | 35.42 (9.75) | 30.06 (10.87)

29. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale at Month 6
Description: as for outcome 28
Time Frame: Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 229 | 216 | 54 | 50
units on a scale | 34.58 (10.69) | 36.30 (10.10) | 33.63 (9.29) | 36.46 (9.27)

30. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score at Baseline and Month 3
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Month 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 240 | 243 | 122
units on a scale
  Baseline (n= 240, 243, 122) | 0.41 (0.32) | 0.39 (0.32) | 0.42 (0.31)
  Month 3 (n= 237, 227, 108) | 0.60 (0.25) | 0.66 (0.23) | 0.51 (0.31)

31. Secondary Outcome: Euro Quality of Life (EQ-5D)- Health State Profile Utility Score at Month 6
Description: as for outcome 30
Time Frame: Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 227 | 214 | 54 | 49
units on a scale | 0.63 (0.23) | 0.68 (0.22) | 0.58 (0.29) | 0.65 (0.21)

32. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Baseline and Month 3
Description: Rheumatoid Arthritis (RA)-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost:visit to doctor,non-medical practitioner,nursing home,hospital,surgery,emergency room(ER) treatment,diagnostic tests, over-night stay,home healthcare services, aids/devices used. Indirect costs associated with functional disability:employment status,willingness to work,work disability due to RA,sick leave,part time work,ability to perform chores,chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale;higher score=higher medical cost.
Time Frame: Baseline, Month 3
Population: FAS population. Participants with at least 1 post-baseline measurement, and baseline measurement for change from baseline endpoint were included. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n'=participants evaluable at given time point for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 236 | 239 | 120
units on a scale
  Baseline:Seen any doctor(n=236,239,119) | 1.19 (0.39) | 1.15 (0.36) | 1.17 (0.38)
  Baseline:Treated in emergency room(n=236,239,120) | 1.94 (0.23) | 1.92 (0.26) | 1.92 (0.28)
  Baseline:Admitted for overnight stay (n=13,18,10) | 0.15 (0.55) | 0.17 (0.51) | 0.20 (0.63)
  Baseline:Hospitalization(n=236,239,120) | 1.94 (0.24) | 1.92 (0.27) | 1.94 (0.24)
  Baseline:Outpatient surgery(n=236,239,120 | 1.97 (0.16) | 1.95 (0.21) | 1.98 (0.16)
  Baseline:Non-study diagnostic test(n=235,239,120) | 1.83 (0.38) | 1.78 (0.41) | 1.83 (0.37)
  Baseline:In nursing home(n=236,239,120) | 1.98 (0.13) | 1.99 (0.09) | 1.99 (0.09)
  Baseline:Home healthcare services(n=235,239,119) | 1.99 (0.09) | 1.98 (0.13) | 1.99 (0.09)
  Baseline:Required aids/devices(n=236,239,119) | 1.84 (0.37) | 1.87 (0.34) | 1.83 (0.38)
  Baseline:Non-medical practitioner(n=236,239,120) | 1.97 (0.18) | 1.99 (0.09) | 1.98 (0.13)
  Baseline:Currently employed(n=236,239,120) | 1.69 (0.46) | 1.64 (0.48) | 1.64 (0.48)
  Baseline:Feel well enough to work(n=111,90,57) | 1.86 (0.35) | 1.83 (0.37) | 1.86 (0.35)
  Baseline:Unable to work due to RA(n=111,93,59) | 1.37 (0.48) | 1.29 (0.46) | 1.41 (0.50)
  Baseline:Lost job/retired early(n=110,92,58) | 1.61 (0.49) | 1.55 (0.50) | 1.55 (0.50)
  Baseline:Work disabled due to RA(n=111,91,58) | 1.54 (0.50) | 1.48 (0.50) | 1.52 (0.50)
  Baseline:Retired(n=116,99,59) | 1.57 (0.50) | 1.57 (0.50) | 1.49 (0.50)
  Baseline:Sick leave due to RA(n=191,202,99) | 1.82 (0.38) | 1.83 (0.38) | 1.74 (0.44)
  Baseline:Performed part time work(n=192,202,98) | 1.89 (0.31) | 1.87 (0.34) | 1.88 (0.33)
  Baseline:Performed paid work(n=191,204,99) | 1.64 (0.48) | 1.66 (0.48) | 1.62 (0.49)
  Baseline:Unable to do chores(n=235,238,118) | 1.36 (0.48) | 1.32 (0.47) | 1.30 (0.46)
  Baseline:Chores by housekeeper(n=235,239,119) | 1.86 (0.35) | 1.82 (0.39) | 1.81 (0.40)
  Baseline:Chores by family/friends(n=235,239,118) | 1.40 (0.49) | 1.44 (0.50) | 1.29 (0.45)
  Month 3:Seen any doctor(n=235,228,109) | 1.42 (0.49) | 1.41 (0.49) | 1.39 (0.49)
  Month 3:Treated in emergency room(n=236,229,109) | 1.94 (0.24) | 1.94 (0.24) | 1.93 (0.26)
  Month 3:Admitted for overnight stay (n=14,14,8) | 0.29 (0.61) | 0.43 (0.65) | 0.50 (0.93)
  Month 3:Hospitalization(n=236,228,109) | 1.99 (0.09) | 1.97 (0.16) | 1.98 (0.13)
  Month 3:Outpatient surgery(n=236,229,109) | 1.97 (0.17) | 1.98 (0.15) | 1.98 (0.13)
  Month 3: Non-study diagnostic test(n=236,228,109) | 1.87 (0.33) | 1.88 (0.32) | 1.87 (0.34)
  Month 3: In nursing home(n=236,229,109) | 2.00 (0.00) | 2.00 (0.07) | 1.99 (0.10)
  Month 3: Home healthcare services(n=236,228,108) | 1.99 (0.09) | 2.00 (0.00) | 1.99 (0.10)
  Month 3: Required aids/devices(n=235,228,109) | 1.89 (0.32) | 1.91 (0.28) | 1.87 (0.34)
  Month 3: Non-medical practitioner(n=236,229,109) | 1.98 (0.13) | 2.00 (0.07) | 2.00 (0.00)
  Month 3: Currently employed(n=236,228,109) | 1.71 (0.45) | 1.65 (0.48) | 1.62 (0.49)
  Month 3: Feel well enough to work(n=108,93,50) | 1.72 (0.45) | 1.69 (0.47) | 1.86 (0.35)
  Month 3: Unable to work due to RA(n=107,98,52) | 1.51 (0.50) | 1.48 (0.50) | 1.35 (0.48)
  Month 3: Lost job/retired early(n=107,92,49) | 1.68 (0.47) | 1.70 (0.46) | 1.59 (0.50)
  Month 3: Work disabled due to RA(n=109,92,49) | 1.57 (0.50) | 1.62 (0.49) | 1.47 (0.50)
  Month 3: Retired(n=115,107,51) | 1.52 (0.50) | 1.51 (0.50) | 1.53 (0.50)
  Month 3: Sick leave due to RA(n=180,183,88) | 1.93 (0.26) | 1.91 (0.29) | 1.89 (0.32)
  Month 3: Performed part time work(n=181,180,88) | 1.94 (0.23) | 1.94 (0.24) | 1.90 (0.30)
  Month 3: Performed paid work(n=179,184,88) | 1.75 (0.44) | 1.76 (0.43) | 1.65 (0.48)
  Month 3: Unable to do chores(n=231,227,107) | 1.60 (0.49) | 1.63 (0.49) | 1.39 (0.49)
  Month 3: Chores by housekeeper(n=235,229,108) | 1.88 (0.32) | 1.92 (0.28) | 1.79 (0.41)
  Month 3: Chores by family/friends(n=234,229,108) | 1.65 (0.48) | 1.64 (0.48) | 1.49 (0.50)

33. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Month 6
Description: as for outcome 32
Time Frame: Month 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 229 | 216 | 54 | 50
units on a scale
  Month 6:Seen any doctor(n=227,216,54,50) | 1.30 (0.46) | 1.30 (0.46) | 1.28 (0.45) | 1.28 (0.45)
  Month 6:Treated in emergency room(n=229,216,54,50) | 1.93 (0.26) | 1.94 (0.24) | 1.94 (0.23) | 1.96 (0.20)
  Month 6:Admitted for overnight stay (n=16,13,3,2) | 0.25 (0.58) | 0.23 (0.44) | 1.33 (2.31) | 1.00 (1.41)
  Month 6:Hospitalization(n=229,216,54,50) | 1.98 (1.15) | 1.99 (1.12) | 1.96 (1.19) | 1.96 (0.20)
  Month 6:Outpatient surgery(n=229,216,54,50) | 1.99 (0.11) | 1.94 (0.23) | 2.00 (0.00) | 1.96 (0.20)
  Month 6:Diagnostic test(n=229,216,54,50) | 1.87 (0.34) | 1.84 (0.37) | 1.87 (0.34) | 1.88 (0.33)
  Month 6:In nursing home(n=229,216,54,50) | 2.00 (0.07) | 2.00 (0.07) | 2.00 (0.00) | 2.00 (0.00)
  Month 6:Home healthcare services(n=229,216,54,49) | 1.99 (0.11) | 2.00 (0.07) | 1.96 (0.19) | 1.98 (0.14)
  Month 6:Required aids/devices(n=229,216,54,50) | 1.89 (0.31) | 1.94 (0.24) | 1.89 (0.32) | 1.92 (0.27)
  Month 6:Non-medical practitioner(n=229,216,54,50) | 2.00 (0.00) | 1.99 (0.10) | 1.98 (0.14) | 2.00 (0.00)
  Month 6:Currently employed(n=229,216,54,50) | 1.71 (0.46) | 1.65 (0.48) | 1.59 (0.50) | 1.58 (0.50)
  Month 6:Feel well enough to work(n=124,101,24,22) | 1.73 (0.45) | 1.66 (0.47) | 1.71 (0.46) | 1.73 (0.46)
  Month 6:Unable to work due to RA(n=123,105,24,24) | 1.50 (0.50) | 1.46 (0.50) | 1.54 (0.51) | 1.42 (0.50)
  Month 6:Lost job/retired early(n=126,102,24,23) | 1.73 (0.45) | 1.63 (0.49) | 1.54 (0.51) | 1.57 (0.51)
  Month 6:Work disabled due to RA(n=125,103,24,23) | 1.62 (0.49) | 1.54 (0.50) | 1.54 (0.51) | 1.43 (0.51)
  Month 6:Retired(n=126,110,25,23) | 1.51 (0.50) | 1.45 (0.50) | 1.56 (0.51) | 1.48 (0.51)
  Month 6:Sick leave due to RA(n=175,169,41,41) | 1.94 (0.23) | 1.94 (0.24) | 1.93 (0.26) | 1.95 (0.22)
  Month 6:Performed part time work(n=173,170,40,41) | 1.93 (0.25) | 1.96 (0.19) | 1.93 (0.27) | 1.95 (0.22)
  Month 6:Performed paid work(n=172,169,39,41) | 1.80 (0.40) | 1.80 (0.40) | 1.64 (0.49) | 1.73 (0.45)
  Month 6:Unable to do chores(n=229,214,52,50) | 1.62 (0.49) | 1.69 (0.46) | 1.54 (0.50) | 1.70 (0.46)
  Month 6:Chores by housekeeper(n=229,216,54,50) | 1.89 (0.31) | 1.94 (0.25) | 1.85 (0.36) | 1.98 (0.14)
  Month 6:Chores by family/friends(n=229,216,54,50) | 1.67 (0.47) | 1.70 (0.46) | 1.54 (0.50) | 1.74 (0.44)

34. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Baseline and Month 3
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA/non-RA related number of visits to doctor, non-medical practitioner, hospital ER treatment, hospitalizations, number of surgeries, diagnostic tests, and devices/aids used were reported.
Time Frame: Baseline, Month 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 193 | 205 | 102
events
  Baseline:Doctor visit(n=193,204,102) | 4.38 (4.50) | 3.85 (4.07) | 3.56 (2.73)
  Baseline:RA related doctor visit (n=192,205,100) | 1.26 (0.81) | 1.18 (0.85) | 1.33 (0.89)
  Baseline:Hospital ER visit(n=13,18,10) | 1.15 (0.38) | 1.61 (1.29) | 1.40 (0.70)
  Baseline:RA related ER visit(n=12,18,10) | 0.75 (0.75) | 0.50 (0.62) | 0.80 (0.92)
  Baseline:Hospitalization(n=14,19,7) | 1.07 (0.27) | 1.11 (0.32) | 1.00 (0.00)
  Baseline:RA related hospitalization(n=14,19,8) | 1.00 (0.55) | 0.84 (0.60) | 0.88 (0.64)
  Baseline:Outpatient surgery(n=6,11,2) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00)
  Baseline:RA related outpatient surgery(n=6,11,3) | 0.00 (0.00) | 0.55 (0.82) | 0.00 (0.00)
  Baseline:Non-study diagnostic test(n=39,51,17) | 1.69 (1.22) | 1.94 (1.22) | 1.59 (1.06)
  Baseline:RA related diagnostic test(n=41,52,19) | 0.61 (0.67) | 0.83 (0.94) | 0.95 (0.97)
  Baseline:Non-medical practitioner visit(n=8,2,2) | 12.00 (12.99) | 7.00 (7.07) | 1.00 (0.00)
  Baseline:RA related non-medical visit(n=8,2,2) | 1.13 (0.64) | 1.50 (0.71) | 0.50 (0.71)
  Month 3:Doctor visit(n=141,137,66) | 3.60 (2.40) | 3.64 (3.44) | 4.00 (3.12)
  Month 3:RA related doctor visit(n=142,138,66) | 0.83 (0.67) | 0.81 (0.81) | 0.92 (0.81)
  Month 3:Hospital ER visit(n=14,14,8) | 1.21 (0.80) | 1.29 (0.47) | 1.50 (0.76)
  Month 3:RA related ER visit(n=14,13,8) | 0.14 (0.53) | 0.15 (0.55) | 0.25 (0.46)
  Month 3:Hospitalization(n=2,6,2) | 1.00 (0.00) | 1.17 (0.41) | 1.00 (0.00)
  Month 3:RA related hospitalization(n=2,7,2) | 0.50 (0.71) | 0.00 (0.00) | 0.00 (0.00)
  Month 3:Outpatient surgery(n=7,5,2) | 1.14 (0.38) | 1.60 (0.89) | 1.00 (0.00)
  Month 3:RA related outpatient surgery(n=7,5,2) | 0.29 (0.76) | 0.00 (0.00) | 1.00 (1.41)
  Month 3:Non-study diagnostic test(n=27,25,13) | 1.26 (0.81) | 1.60 (0.82) | 1.54 (0.78)
  Month 3:RA related diagnostic test(n=30,26,14) | 0.13 (0.35) | 0.15 (0.37) | 0.21 (0.43)
  Month 3:Non-medical practitioner visit(n=4,1,0) | 10.75 (6.99) | 7.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Month 3:RA related non-medical visit(n=4,1,0) | 0.25 (0.50) | 2.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.

35. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Month 6
Description: as for outcome 34
Time Frame: Month 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 159 | 152 | 39 | 36
events
  Doctor visit(n=159,152,39,36) | 3.22 (2.54) | 3.69 (3.18) | 3.00 (2.29) | 3.69 (2.25)
  RA related doctor visit(n=159,152,39,36) | 0.92 (0.70) | 0.83 (0.73) | 1.05 (0.60) | 0.92 (0.69)
  Hospital ER visit(n=16,13,3,2) | 1.06 (0.25) | 1.25 (0.45) | 3.00 (1.73) | 1.00 (0.00)
  RA related ER visit(n=16,12,3,2) | 0.13 (0.34) | 0.08 (0.28) | 1.67 (2.08) | 0.00 (0.00)
  Hospitalization(n=5,3,2,2) | 1.20 (0.45) | 1.00 (0.00) | 1.50 (0.71) | 1.00 (0.00)
  RA related hospitalization(n=5,3,2,2) | 0.20 (0.45) | 0.33 (0.58) | 0.50 (0.71) | 0.00 (0.00)
  Outpatient surgery(n=3,10,0,2) | 1.00 (0.00) | 1.50 (1.58) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 1.00 (0.00)
  RA related outpatient surgery(n=3,12,0,2) | 0.00 (0.00) | 0.00 (0.00) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 0.00 (0.00)
  Non-study diagnostic test(n=24,33,7,5) | 2.04 (1.55) | 1.39 (0.75) | 2.57 (1.62) | 1.20 (0.45)
  RA related diagnostic test(n=29,34,6,6) | 0.45 (0.87) | 0.29 (0.52) | 0.67 (0.82) | 0.33 (0.52)
  Non-medical practitioner visit(n=0,2,0,0) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 3.00 (1.41) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  RA related non-medical visit(n=0,2,0,0) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 0.50 (0.71) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.

36. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Baseline and Month 3
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains.Any RA or non-RA related number of days spent in hospital, nursing home, aids/devices used, on sick leave, work per week, performed part time work, performed paid work, chores done by housekeeper and chores done by family/friends.
Time Frame: Baseline, Month 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 139 | 131 | 84
days
  Baseline:Hospital length of stay(n=14,19,7) | 15.43 (12.33) | 9.63 (7.27) | 4.29 (2.81)
  Baseline:Days in nursing home(n=4,2,1) | 23.25 (2.63) | 16.50 (6.36) | 10.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Baseline:Days devices/aids used(n=37,31,20) | 118.95 (134.74) | 85.52 (95.38) | 55.90 (56.66)
  Baseline:RA related aids used(n=38,31,20) | 2.21 (1.47) | 1.90 (1.33) | 1.45 (0.69)
  Baseline:Days of work per week(n=72,84,43) | 5.08 (1.04) | 4.92 (1.17) | 5.02 (0.96)
  Baseline:Days on sick leave(n=33,34,25) | 25.12 (33.23) | 10.91 (18.15) | 22.40 (29.72)
  Baseline:Days of part time work(n=20,25,12) | 15.65 (22.74) | 20.44 (26.71) | 12.42 (10.57)
  Baseline:Paid work, bothered by RA(n=69,68,37) | 33.87 (31.01) | 28.15 (29.06) | 38.30 (27.52)
  Baseline:Chores by housekeeper(n=33,43,22) | 17.30 (24.67) | 16.63 (25.99) | 14.55 (22.32)
  Baseline:Chores by family(n=139,131,84) | 29.54 (31.72) | 27.85 (34.80) | 22.12 (27.36)
  Month 3:Hospital length of stay(n=2,6,2) | 7.50 (6.36) | 6.33 (7.12) | 12.00 (2.83)
  Month 3:Days in nursing home(n=0,1,1) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 2.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 10.0 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 3:Days devices/aids used(n=27,20,14) | 109.93 (107.85) | 89.50 (89.98) | 94.68 (111.05)
  Month 3:RA related aids used(n=27,20,14) | 1.81 (1.36) | 1.50 (0.95) | 1.93 (1.21)
  Month 3:Days of work per week(n=68,79,41) | 5.00 (0.93) | 5.05 (1.19) | 4.88 (1.17)
  Month 3:Days on sick leave(n=13,17,10) | 15.00 (23.59) | 14.82 (23.32) | 19.60 (27.68)
  Month 3:Days of part time work(n=10,11,9) | 12.70 (20.97) | 19.09 (25.07) | 6.22 (5.70)
  Month 3:Paid work, bothered by RA(n=44,44,30) | 21.70 (26.22) | 19.39 (23.10) | 26.50 (27.03)
  Month 3:Chores by housekeeper(n=26,19,23) | 7.73 (8.43) | 6.32 (5.73) | 18.13 (25.19)
  Month 3:Chores by family(n=81,82,55) | 25.72 (31.12) | 27.29 (33.02) | 27.00 (30.37)

37. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Month 6
Description: as for outcome 36
Time Frame: Month 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 74 | 75 | 24 | 21
days
  Hospital length of stay(n=5,3,2,2) | 13.60 (18.28) | 7.67 (5.86) | 13.50 (14.85) | 1.50 (0.71)
  Days in nursing home(n=1,1,0,0) | 24.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 15.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter.
  Days devices/aids used(n=24,13,6,4) | 97.17 (116.84) | 53.85 (52.29) | 101.50 (106.85) | 72.25 (113.10)
  RA related aids used(n=25,12,6,4) | 1.48 (1.23) | 1.67 (0.98) | 2.17 (1.83) | 1.75 (0.96)
  Days of work per week(n=65,75,22,21) | 4.95 (0.84) | 5.16 (0.99) | 5.09 (1.15) | 4.71 (1.19)
  Days on sick leave(n=10,10,3,2) | 21.10 (27.23) | 15.50 (27.71) | 9.00 (5.20) | 47.50 (60.10)
  Days of part time work(n=11,6,3,2) | 15.00 (25.46) | 8.50 (5.68) | 5.00 (3.00) | 4.00 (4.24)
  Paid work, bothered by RA(n=34,32,14,12) | 21.09 (25.89) | 12.72 (17.50) | 26.14 (29.98) | 15.92 (18.80)
  Chores by housekeeper(n=25,13,8,1) | 16.32 (24.40) | 20.23 (31.76) | 8.50 (11.78) | 90.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Chores by family(n=74,64,24,13) | 20.38 (27.42) | 28.09 (32.55) | 11.58 (18.35) | 27.38 (30.61)

38. Secondary Outcome: Number of Hours Per Day as Assessed RA-HCRU at Baseline and Month 3
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of hours spent per day for home healthcare services, chores done by housekeeper, chores done by family or friends, work done and work missed were reported.
Time Frame: Baseline, Month 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 139 | 131 | 82
hours per day
  Baseline:Home healthcare services(n=1,4,1) | 2.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 3.75 (5.50) | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Baseline:RA related home HC services(n=2,4,1) | 1.50 (0.71) | 2.25 (2.50) | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Baseline:Work done(n=71,85,43) | 7.66 (1.87) | 8.60 (6.12) | 8.95 (5.20)
  Baseline:Missed work due to RA(n=19,25,12) | 3.47 (2.67) | 10.84 (24.54) | 6.17 (12.29)
  Baseline:Chores by housekeeper(n=33,43,22) | 5.64 (4.06) | 4.67 (2.07) | 5.86 (3.06)
  Baseline:Chores by family(n=139,131,82) | 3.99 (4.02) | 3.32 (2.89) | 4.85 (6.88)
  Month 3:Home healthcare services(n=2,0,1) | 2.50 (2.12) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 3:RA related home HC services(n=2,0,1) | 0.50 (0.71) | NA (NA) — Data was not analyzed as no participant was evaluable for this parameter. | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Month 3:Work done(n=66,79,41) | 8.20 (7.28) | 7.68 (2.37) | 8.85 (5.34)
  Month 3:Missed work due to RA(n=10,9,9) | 2.20 (1.55) | 3.67 (1.41) | 9.56 (19.04)
  Month 3:Chores by housekeeper(n=27,19,23) | 5.74 (4.70) | 5.21 (4.89) | 5.91 (4.75)
  Month 3:Chores by family(n=79,82,54) | 3.09 (1.96) | 3.82 (6.91) | 3.69 (3.82)

39. Secondary Outcome: Number of Hours Per Days as Assessed Using RA-HCRU at Month 6
Description: as for outcome 38
Time Frame: Month 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 74 | 75 | 24 | 21
hours per day
  Home healthcare services(n=3,1,1,1) | 4.00 (1.00) | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  RA related home healthcare services(3,1,2,1) | 1.00 (1.00) | 1.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 0.00 (0.00) | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Work done(n=65,75,22,21) | 8.38 (5.53) | 8.43 (4.16) | 7.23 (2.11) | 8.29 (1.79)
  Missed work due to RA(n=11,7,3,2) | 2.73 (2.53) | 2.57 (1.72) | 2.67 (2.31) | 1.50 (2.12)
  Chores by housekeeper(n=24,14,8,1) | 5.13 (2.49) | 10.57 (22.97) | 5.00 (2.45) | 8.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.
  Chores by family(n=74,64,24,13) | 3.11 (2.18) | 2.86 (1.80) | 3.29 (2.84) | 4.69 (6.46)

40. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU at Baseline and Month 3
Description: Work performance of participants on number of days bothered was based on a 0 to 10-point scale, where higher score indicated lower work performance.
Time Frame: Baseline, Month 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 148 | 174 | 79
units on a scale
  Baseline (n=146, 174, 79) | 5.59 (3.17) | 5.61 (6.42) | 5.41 (2.94)
  Month 3 (n=138, 148, 75) | 3.39 (2.85) | 3.43 (2.88) | 4.57 (2.94)

41. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU at Month 6
Description: as for outcome 40
Time Frame: Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 130 | 138 | 34 | 34
units on a scale | 3.22 (2.85) | 3.18 (3.00) | 3.21 (2.80) | 3.94 (3.22)

42. Other Pre Specified Outcome: Time to First Greater Than 1 Day Sequential Decrease in Pain From Baseline for Patient Assessment of Arthritis Pain
Description: as for outcome 16
Time Frame: 2 weeks
Population: as for outcome 3
Measure: Number; unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 59 | 61 | 31
days | 3 | 3 | 3

43. Other Pre Specified Outcome: Time to First Greater Than 1 Day Sequential Decrease in Pain From Baseline for Patient Global Assessment of Arthritis
Description: as for outcome 18
Time Frame: 2 weeks
Population: as for outcome 3
Measure: Number; unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 59 | 61 | 31
days | 3 | 3 | 3

44. Secondary Outcome: Work Limitations Questionnaire (WLQ) Score at Baseline and Month 3
Description: WLQ: participant-reported 25-item scale to evaluate degree to which health problems interfere with an ability to perform job roles along 4 dimensions: Time Management scale (5-items); Physical Demands scale (6-item); Mental-Interpersonal Demands Scale (9-items); Output Demands scale (5-items). All the scales ranged from 0 (limited none of the time) to 100 (limited all of the time). Work Loss Index, which represented percentage of lost work over time period relative to a normative population, was derived (total score:0[no loss] to 100[complete loss of work]).
Time Frame: Baseline, Month 3
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo
Number analyzed (Participants) | 124 | 122 | 67
units on a scale
  Baseline:Time management(n=118, 119, 62) | 50.84 (26.52) | 48.98 (27.17) | 48.74 (26.44)
  Baseline:Physical demands(n=117, 119, 66) | 51.84 (22.44) | 49.24 (27.51) | 51.21 (25.33)
  Baseline:Mental demands(n=119,120,66) | 31.04 (24.05) | 36.14 (28.41) | 38.69 (27.76)
  Baseline:Output demands(n=114, 116, 63) | 39.70 (24.76) | 44.85 (30.23) | 45.30 (28.11)
  Baseline:Work loss index(n=124, 122, 67) | 10.82 (5.21) | 11.95 (6.20) | 12.16 (5.92)
  Month 3:Time management(n=94, 89, 45) | 37.65 (29.03) | 34.63 (29.91) | 41.32 (23.28)
  Month 3:Physical demands(n=98, 90, 46) | 51.89 (29.32) | 46.48 (30.17) | 46.71 (24.78)
  Month 3:Mental demands(n=100, 93, 47) | 24.64 (27.02) | 24.62 (29.12) | 28.54 (26.40)
  Month 3:Output demands(n=96, 90, 45) | 27.03 (24.44) | 28.31 (29.37) | 33.41 (23.28)
  Month 3:Work loss index(n=102, 98, 49) | 8.48 (5.60) | 8.05 (6.63) | 9.29 (5.66)

45. Secondary Outcome: Work Limitations Questionnaire (WLQ) Score at Month 6
Description: as for outcome 44
Time Frame: Month 6
Population: FAS population. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n'=participants evaluable at given parameter for each group respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg
Number analyzed (Participants) | 85 | 85 | 26 | 27
units on a scale
  Time management (n=80, 81, 25, 23) | 36.27 (29.22) | 30.42 (28.39) | 34.40 (25.59) | 39.86 (30.64)
  Physical demands (n=85, 81, 26, 25) | 45.37 (29.86) | 45.17 (34.14) | 57.16 (27.63) | 50.33 (31.74)
  Mental demands (n= 81, 82, 25, 26) | 22.66 (25.71) | 21.61 (29.09) | 25.84 (24.54) | 29.77 (29.64)
  Output demands (n= 80, 81, 26, 23) | 25.04 (24.29) | 26.30 (29.40) | 28.65 (23.90) | 35.05 (29.32)
  Work loss index (n= 85, 85, 26, 27) | 7.85 (5.64) | 7.60 (6.49) | 9.07 (5.22) | 9.23 (6.26)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- CP-690550 5 mg (Up To Month 3): CP-690550 5 mg tablet orally twice daily up to Month 3.
- CP-690550 10 mg (Up To Month 3): CP-690550 10 mg tablet orally twice daily up to Month 3.
- Placebo (Up To Month 3): Matching placebo tablet orally twice daily up to Month 3.
- CP-690550 5 mg (Post Month 3): CP-690550 5 mg tablet orally twice daily from Month 3 to Month 6.
- CP-690550 10 mg (Post Month 3): CP-690550 10 mg tablet orally twice daily from Month 3 to Month 6.
Arm/Group | CP-690550 5 mg (Up To Month 3) | CP-690550 10 mg (Up To Month 3) | Placebo (Up To Month 3) | CP-690550 5 mg (Post Month 3) | CP-690550 10 mg (Post Month 3)
Serious Adverse Events (participants affected / at risk) | 1/243 | 5/245 | 6/122 | 6/304 | 6/306
Other Adverse Events (participants affected / at risk) | 80/243 | 84/245 | 40/122 | 37/304 | 48/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690550 5 mg (Up To Month 3) (N=243) | CP-690550 10 mg (Up To Month 3) (N=245) | Placebo (Up To Month 3) (N=122) | CP-690550 5 mg (Post Month 3) (N=304) | CP-690550 10 mg (Post Month 3) (N=306)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominoplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Breast prosthesis implantation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690550 5 mg (Up To Month 3) (N=243) | CP-690550 10 mg (Up To Month 3) (N=245) | Placebo (Up To Month 3) (N=122) | CP-690550 5 mg (Post Month 3) (N=304) | CP-690550 10 mg (Post Month 3) (N=306)
Anaemia (Blood and lymphatic system disorders) | 4 | 6 | 2 | 3 | 7
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 5 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 9 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 6 | 4 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 6 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 9 | 3 | 0 | 0
Oedema peripheral (General disorders) | 7 | 5 | 3 | 1 | 7
Pyrexia (General disorders) | 2 | 1 | 3 | 0 | 0
Influenza (Infections and infestations) | 2 | 4 | 4 | 5 | 6
Nasopharyngitis (Infections and infestations) | 4 | 5 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 8 | 6 | 14 | 8
Urinary tract infection (Infections and infestations) | 4 | 10 | 3 | 3 | 11
Blood creatine phosphokinase increased (Investigations) | 3 | 10 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 2 | 1 | 8
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 5 | 4 | 0 | 0
Headache (Nervous system disorders) | 13 | 11 | 3 | 9 | 7
Paraesthesia (Nervous system disorders) | 6 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 7 | 2 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.